CLINICAL TRIAL: NCT06454006
Title: Effects of Photobiomodulation Therapy Combined With Static Magnetic Field in Reducing the Number of Days in the Intensive Care Unit (ICU) for Adult Patients Requiring Mechanical Ventilation
Brief Title: Effects of PBMT-sMF in Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6.738.501
Record Dates: First submitted 2024-05-28; First posted 2024-06-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Failure
Keywords: Mechanical ventilation; Photobiomodulation therapy; LLLT; Static magnetic field; Diaphragm; Intensive care unit
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (placebo or active) and will be instructed not to inform the patients, therapists or other researchers as to the type of treatment (placebo or active). Therefore, the patients, therapists, and the outcome assessors will be blinded to the type of treatment being administered to the patients. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (placebo or active).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment will be delivered using Multi Radiance® Medical PhotOxyl photoceutical medical device emitting a light source that is sufficient to be indistinguishable from the active comparator but does not deliver any therapeutic energy, combined with standard of care therapy for a mechanically ventilated patient in the ICU.
  The treatment administration protocol comprises one 7-minute treatment administration per day on each consecutive day for four consecutive weeks, for a maximum of 28 consecutive treatments over 28 consecutive days, or until the day of the subject's successful weaning from mechanical ventilation, or until the day of the subject's death, whichever occurs first.
  Interventions: Device: Placebo PBMT-sMF
- Active (Active Comparator): Active treatment will be delivered using Multi Radiance® Medical PhotOxyl photoceutical medical device in active mode, combined with standard of care therapy for a mechanically ventilated patient in the ICU.
  The treatment administration protocol comprises one 7-minute treatment administration per day on each consecutive day for four consecutive weeks, for a maximum of 28 consecutive treatments over 28 consecutive days, or until the day of the subject's successful weaning from mechanical ventilation, or until the day of the subject's death, whichever occurs first.
  Interventions: Device: Active PBMT-sMF

INTERVENTIONS:
Device: Placebo PBMT-sMF — Placebo, without therapeutic dose.
  Arms: Placebo
Device: Active PBMT-sMF — Active with a dose of 31.50 J per site.
  Arms: Active

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of photobiomodulation therapy combined with static magnetic field (PBMT-sMF) in adult patients who require mechanical ventilation. The main questions it aims to answer are:

(i) Does PBMT-sMF lower the length of stay in the intensive care unit (ICU) for mechanically ventilated patients? (ii) Does PBMT-sMF increase the diaphragm thickness in mechanically ventilated patients in the ICU?

Researches will compare active PBMT-sMF plus standard of care to a placebo PBMT-sMF plus standard of care to see if active PBMT-sMF works to prevent or retard disuse atrophy of the diaphragm during mechanical ventilation.

DETAILED DESCRIPTION:
To achieve the proposed objectives it will be performed a multi-center, randomized, triple-blinded (patients, therapists, outcome assessors), placebo-controlled trial, in patients who required mechanical ventilation.

One hundred and twelve patients will be randomly allocated to two treatment groups:

1. Active treatment: Patients will receive treatment with the active PBMT-sMF combined with standard of care therapy for a mechanically ventilated patient in the ICU.
2. Placebo treatment: Patients will receive treatment with the placebo PBMT-sMF combined with standard of care therapy for a mechanically ventilated patient in the ICU.

The randomization will occur immediately following patients qualification and prior to any additional study activities occurring.

The treatment administration protocol (28-day administration protocol) will comprise: 7-minute treatment administration per day on each consecutive day for four consecutive weeks, for a maximum of 28 consecutive treatments over 28 consecutive days, or until the day of the patient's successful weaning from mechanical ventilation, or until the day of the patient's death, whichever occurs first.

The data will be collected by a blinded assessor.

Due to the nature of the condition being evaluated in this study, the study assessment timeline is patient dependent and will therefore be unique to each patient.

The study will comprise:

1. pre-treatment evaluation phase (before starting treatment);
2. treatment administration phase (two assessments: after completion of 14 and 28 days of treatment);
3. post-treatment evaluation phase (any patient who is not discharged from the hospital or who does not die during the treatment administration and evaluation phase will proceed to the post-treatment administration phase. The post-treatment phase will start on the day immediately following the patient's last day in the treatment administration evaluation phase. The post-treatment phase will end on the day that the patient is discharged from the hospital, or the day that the patient dies prior to discharge from the hospital, whichever occurs firs. Therefore, the duration of the post-treatment administration phase will vary by individual patient. During the post-treatment evaluation period, the following assessments will be recorded once every two weeks, as applicable, with the final post-treatment evaluation visit determined on an individual patient basis, up to 2 years).

P.S.:

* For patients whose successful weaning from mechanical ventilation occurs prior to completion of the 28-day administration protocol, the endpoint assessment visit will occur on or after the day of successful weaning.
* For patients who die before completion of the 28-day administration protocol, the endpoint assessment visit will include outcome measures recorded as close to the date of the patient's death as possible.

The investigators will analyze: 1) Length of stay in the ICU; 2) Diaphragm thickness; 3) Length of stay in the hospital following ICU discharge; 4) Length of time until weaning from mechanical ventilation; 5) Mechanical ventilation parameters: (i) Positive end-expiratory pressure levels (PEEP) and (ii) Fraction of inspired oxygen (FiO2); 6) Arterial blood gas analysis: (i) Arterial partial pressure of oxygen (PO2) and (ii)PO2/FiO2 ratio; 7) Vital signs: blood pressure, heart rate, SpO2, blood glucose, etc.; 8) Blood draw analysis: C-reactive protein (CRP); Tumor necrosis factor-alpha (TNF-α); Vitamin D; erythrocytes; hemoglobin; hematocrit; leucocytes; segmented neutrals; eosinophiles; basophiles; lymphocytes; monocytes; platelet count;8) Survival rate; 9) Local skin reactions; 10) Adverse events and serious adverse events.

The statistical analysis will follow the intention-to-treat principles.

ELIGIBILITY:
Inclusion Criteria:

* Legally authorized representative signed informed consent;
* Male or female aged 21 years or older;
* On mechanical ventilation through orotracheal intubation for no more than 72 hours prior to study enrollment or pending mechanical ventilation through orotracheal intubation;
* Predicted to remain on mechanical ventilation for at least 48 hours (≥48 hours) from the time of study enrollment

Exclusion Criteria:

* Mechanical ventilation initiated longer than 72 hours prior to anticipated enrollment;
* Body Mass Index (BMI) > 40 kg/m²;
* Fever of 100.4°C or higher;
* Situated in the prone position for 24 hours or longer during mechanical ventilation;
* Prognosis of mortality within 72 hours, per the patient's physician;
* Hypersensitivity to light;
* Use of non-invasive ventilation, Continuous Positive Airway Pressure (CPAP) and/or Bilevel Positive Airway Pressure (BiPAP) device for ≥ 50% of the time over the preceding 6 months;
* Tracheostomy;
* Any one or more of the following present on both sides of the neck (bilaterally) at the intended treatment site(s): internal jugular (IJ) venous cannulation; incisions, significant bruising; burn(s); notable skin irritation/rash, or other skin condition that may place the subject at risk from harm from the device treatment;
* Fracture, external or internal hemorrhage, or at risk of hemorrhage following acute trauma or fracture, or known or potential acute occult bleeding (e.g., gastric ulcer, intestine) in the intended treatment areas;
* Metallic device implants or body penetrating metallic devices in the upper body/neck area whose location may interfere with the study device treatment administration. E.g., extracorporeal membrane oxygenation (ECMO) cannula;
* Non-removable electrical/electronic device in the upper body/neck area that may interfere with the study device treatment administration, e.g., -implanted pacemaker or cardiac defibrillator;
* Cardiogenic or septic shock with ongoing severe hemodynamic instability (according to the American College of Chest Physicians definition (that cannot be stabilized within the 48 hours enrollment period);
* Conditions that may limit ultrasonographic assessment of diaphragmatic thickness, e.g., occluding chest drain, pleural effusion, pulmonary consolidation of the lower lobe(s);
* Current cancer of any type;
* Pregnancy;
* Any comorbidity, co-existing condition or illness, or other factor that in the opinion of the study investigator may render the subject unsuitable for participation in the study;
* Admission to the ICU within the last 12 months due to respiratory distress/failure;
* Two or more admissions to the ICU within the prior 12 months for any reason;
* Current participation in another clinical study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Length of stay in the intensive care unit (ICU) | From date of ICU admission until the date of discharge or date of death from any cause, whichever came first, assessed up to 28 days.
  Number of days hospitalized in the ICU until discharge from ICU or death from any cause.

SECONDARY OUTCOMES:
Length of stay in the hospital | Assessments once every two weeks after discharge from ICU until the date of discharge of hospital or date of death from any cause, whichever came first, up to 2 years.
  Number of days from the patient's admission to the hospital, following discharge from the ICU, to the patient's discharge from the hospital or death from any cause, whichever came first.
Length of time until weaning from mechanical ventilation (MV) | After 14 days of treatment; after 28 days of treatment; and once every two weeks until the date of successful weaning from MV or date of death, whichever came first, up to 2 years.
  The number of days from patient initiation on MV until successful weaning.
Levels of positive end-expiratory pressure levels (PEEP) | After 14 days of treatment; after 28 days of treatment; and once every two weeks until the date of successful weaning from MV or date of death, whichever came first, up to 2 years.
  The levels of PEEP will be measured using a mechanical ventilator.
Levels of fraction of inspired oxygen (FiO2) | After 14 days of treatment; after 28 days of treatment; and once every two weeks until the date of successful weaning from MV or date of death, whichever came first, up to 2 years.
  The levels of PEEP will be measured using a mechanical ventilator.
Arterial partial pressure of oxygen (PO2) | After completion of 14 days of treatment; after completion of 28 days of treatment, and assessments once every two weeks until the date of successful weaning from mechanical ventilation or date of death, whichever came first, up to 2 years.
  PO2 will be measured by arterial blood gas analysis.
Arterial partial pressure of oxygen (PO2)/Fraction of inspired oxygen (FiO2) ratio | After 14 days of treatment; after 28 days of treatment; and once every two weeks until the date of successful weaning from MV or date of death, whichever came first, up to 2 years.
  PO2 will be measured by arterial blood gas analysis.
C-reactive protein (CRP) | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  CRP will be measured by blood test.
Erythrocytes | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Erythrocytes will be measured by blood test.
Hemoglobin | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Hemoglobin will be measured by blood test.
Hematocrit | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Hematocrit will be measured by blood test.
Leucocytes | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Leucocytes will be measured by blood test.
Segmented neutrals | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Segmented neutrals will be measured by blood test.
Eeosinophiles | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Eosinophiles will be measured by blood test.
Basophiles | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Basophiles will be measured by blood test.
Lymphocytes | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Lymphocytes will be measured by blood test.
Monocytes | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Monocytes will be measured by blood test.
Platelet count | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Platelet count will be measured by blood test.
Survival rate | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Rate of how many people survived and were discharged and how many died.
Local skin reactions | After each treatment administration up to 28 days.
  Local skin reaction will be measured by four-point post-treatment assessment severity scale
Adverse events | Adverse events will be collected throughout study duration up to 2 years.
  All adverse events that occur after randomization, including local and systemic reactions, not meeting the criteria for serious adverse events will be captured on the appropriate adverse event case report form.
End-expiratory diaphragm thickness | After 14 days of treatment; after 28 days of treatment; and once every two weeks after discharge from ICU until the date of discharge of hospital or death from any cause, whichever came first, up to 2 years.
  Diaphragm thickness will be measured by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during five years after the study completion.
Access Criteria: All IPD that underlie results in a publication will be available on reasonable request.